CLINICAL TRIAL: NCT03093363
Title: Study of the Impact of a Hospital Pharmacist's Intervention in Collaboration With Pneumologists on Bronchial Inflammation of Outpatient Asthmatic Patients Seen in University Hospital of Liege
Brief Title: Impact of a Hospital Pharmacist's Intervention on FENO (Fractional Exhaled Nitric Oxide) in Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Renaud Louis, Professor, MD, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B707201629850
Record Dates: First submitted 2017-03-11; First posted 2017-03-28 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Asthmatic patients with the pharmacist's intervention
  Interventions: Other: Pharmacist's intervention
- Control group (Other): Asthmatic patients without the pharmacist's intervention (only questionnaires)
  Interventions: Other: Questionnaires for control group

INTERVENTIONS:
Other: Pharmacist's intervention — Pharmacist's intervention with asthmatic patients:
  * Detailed questionnaire on asthma and treatments (atopy, comorbidities, smoking status, asthma control, adverse effects of treatments, etc.)
  * Explanation of asthma and inflammation
  * Explanation of triggers and how to avoid it
  * Explanation of asthma treatments
  * Explanation of the inhalation technique with a physical demonstration
  * Emphasis on treatment adherence
  * Assessment of comorbidities and their treatment
  * Emphasis on influenza vaccination
  Arms: Intervention group
Other: Questionnaires for control group — - Detailed questionnaire on asthma and treatments (atopy, comorbidities, smoking status, asthma control, adverse effects of treatments, etc.)
  Arms: Control group

SUMMARY:
The impact of a pharmacist's intervention on asthma control has now been well demonstrated, but its effect on inflammatory markers of FENO (Fractional exhaled nitric oxide) in asthmatic patients has been little studied in the literature. The aim of this study is to investigate the impact of a pharmacist's intervention on FENO in patients seen in clinical practice by a pneumologist in a secondary university center.

ELIGIBILITY:
Inclusion Criteria:

* Adult asthmatics (definition of asthma: FEV1 [forced expiratory volume in 1 second] reversibility of at least 12% and 200 mL after 400 mcg of salbutamol and/or PC20M [provocative concentration of methacholine causing a 20% fall in FEV1]<16 mg/mL)
* unchanged or increased dose of inhaled corticosteroids prescribed by the pneumologist at the visit
* FENO (fractional exhaled nitric oxide) > or = 25 ppb

Exclusion Criteria:

* Treatment with oral corticosteroids to treat an asthma exacerbation within 4 weeks before the visit with the pneumologist

Exclusion Criteria during the study:

* Change of the dose of ICS (inhaled corticosteroids) during the follow-up of 3 months after the pharmacist's intervention
* Severe asthma exacerbation requiring oral corticosteroids within the 4 weeks before the follow-up visit (3 months after the pharmacist's intervention)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline FENO (fractional exhaled nitric oxide) at 3 months | 3 months
  Fractional exhaled nitric oxide

SECONDARY OUTCOMES:
Change from Baseline FEV1 (forced expiratory volume in 1 second) at 3 months | 3 months
Change from Baseline FVC (forced vital capacity) at 3 months | 3 months
Change from Baseline FEV1/FVC at 3 months | 3 months
Change from Baseline ACQ (Asthma Control Questionnaire) at 3 months | 3 months
Change from Baseline ACT (Asthma Control Test) at 3 months | 3 months
Change from Baseline miniAQLQ (Asthma Quality of Life Questionnaire) at 3 months | 3 months
Change from Baseline MARS (Medication Adherence Report Scale) at 3 months | 3 months
  Measure of treatment adherence
Change from Baseline MRA (Medication Refill Adherence) at 3 months | 3 months
  Measure of treatment adherence
Change from Baseline score of the inhalation technique at 3 months | 3 months
Change from Baseline number of severe exacerbations (during the 3 previous months) at 3 months | 3 months
  Severe exacerbations are asthma exacerbations requiring oral corticosteroids
Change from Baseline smoking status at 3 months | 3 months
  Smoking status is recorded as non-smoker, ex-smoker, current smoker
Satisfaction of patients with the pharmacist's intervention, with a scale from 0 to 10 | 3 months after intervention
Changes in lifestyle related to asthma (free text field to complete by the patient) | 3 months after intervention

IPD SHARING:
Plan to Share IPD: Undecided